CLINICAL TRIAL: NCT02606578
Title: Achalasia Patient Reported Outcomes
Status: Terminated | Type: Observational
Why Stopped: Study's original Principal Investigator no longer at the institution.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Janani S. Reisenauer, Principal Investigator, Mayo Clinic
Other Study IDs: 15-006921
Record Dates: First submitted 2015-11-09; First posted 2015-11-17 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Achalasia; Achalasia; Achalasia, Esophageal
MeSH Terms: conditions — Esophageal Achalasia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Questionnaires — The study team will collect information from your medical record regarding: demographics, operation, nutritional status, laboratory values, testing results, complications, hospital data, cost, length of stay, past medical history and clinical outcomes.
  At your clinical follow-up visits (~4 weeks, 6 months, and 12 months post operation), a study coordinator will meet with you to assess for adverse events and to have you complete research questionnaires. Alternatively, the study coordinator may call you to assess for adverse events and ask if we can mail you the research questionnaires to complete and mail back.
  You will also be asked to complete the research questionnaires a minimum of once a year for your lifetime: A study coordinator will call you and ask if we can mail you questionnaires to complete and mail back.

SUMMARY:
Patients that are either scheduled to undergo or have undergone an achalasia procedure at the Mayo Clinic Rochester are asked to participate. The purpose of this study is to gather information and determine if one of these procedures is superior to the other.

DETAILED DESCRIPTION:
This is a non-randomized, non-inferiority trial that has been created to compare results of achalasia procedures including but not limited to: POEM + Partial Fundoplication (PF), POEM and Laparoscopic Modified Heller Myotomy + PF and POEM + Peroral Plication of the esophagus. Using a set of consistent evaluation tools for patients undergoing treatment for achalasia allows a standardized evaluation and comparison of these groups of patients. The long term and comparative POEM procedure outcomes are not currently known. Patients undergoing POEM, fundoplication, and/or laparoscopic myotomy report having varying degrees of symptoms of reflux, dysphagia, and pain. Providers also note varying degrees of esophagitis by endoscopy, reflux by impedance or pH scoring, and recurrence by repeat manometry. Many of these issues can be quantified using pH probe testing, upper GI endoscopy, high resolution manometry, CT scans, Endoflip device and esophagrams. There are various validated questionnaires that have been used to assess problem areas of reflux, dysphagia, and pain such as the Promis Global Health Score, Ekhardt Score, Mayo GER Score, Modified Dysphagia Questionnaire-30 Day, Zubrod Score, and pain scale. Each of these symptoms, tests, and questionnaires contributes to the provider's understanding of the patient's postoperative outcome.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Undergoing a POEM or laparoscopic modified heller myotomy and anti-reflux procedures
* Esophagus diameter less <8 cm on barium swallow test

Exclusion Criteria:

* Pregnant
* Diverticular disease of the esophagus
* Barrett's esophagus
* Extensive abdominal adhesions
* <50% predicted FEV1 on pulmonary function testing
* Cardiac ejection fraction <25%
* Esophageal stricture from prior myotomy
* Sigmoidization of the esophagus
* More than one prior balloon dilation (>3 cm) or any prior dilation of 3 cm

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing PerOral Endoscopic Myotomy (POEM) or Laparoscopic Modified Heller Myotomy and Anti-Reflux Procedures at Mayo Clinic Rochester
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-10; Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Comparison of different surgical techniques with patient reported post-operative symptoms on the achalasia questionnaire | 2 years
  Comparison of surgical techniques evaluated from the patient's medical record using patient reported post-operative symptoms on the achalasia questionnaire. The achalasia questionnaire includes quality of life, pain, activity level, heart burn, acid regurgitation, reflux, dysphagia, and diet.

CONTACTS AND LOCATIONS:
Overall Officials: Janani Reisenauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials